CLINICAL TRIAL: NCT04267783
Title: Prediction of Uterine Atony After Vaginal Delivery by Shear Wave Elastography: a Feasibility Study
Brief Title: Prediction of Uterine Atony After Vaginal Delivery by Elastography
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, DAVID DESSEAUVE, Principal investigator, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 2018-02267
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Postpartum Hemorrhage
Keywords: postpartum hemorrhage; uterine atony; shear wave; elastography
MeSH Terms: conditions — Postpartum Hemorrhage; Uterine Inertia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Shear wave elastography — Investigate the feasibility of use of shear-wave elastography of the uterus during the third stage of labour and following placental delivery in order to predict uterine atony .

SUMMARY:
Prospective study evaluating the feasibility of shear-wave elastography of the uterus during the third stage of labour and following placental delivery. The investigators hypothesize that the stiffness of the myometrium can be measured by using shear-wave technology. This study involves 30 patients with a healthy pregnancy and spontaneous vaginal delivery. One co-investigator will carry out measurements at the uterine fundus, at three different time points: after fetal delivery, after placental delivery and 30 minutes after placental delivery.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* cephalic presentation
* maternal age > 18 years old
* nulliparous
* healthy uncomplicated pregnancy
* gestational age between 37-42 weeks of gestation
* spontaneous labour and delivery
* uncomplicated progression of labour (cervical dilatation at >1 cm/h)
* administration of less than 3 units of oxytocin during the second stage of labour
* patient having read, accepted and signed the consent form

Exclusion Criteria:

* antepartum hemorrhage in the present pregnancy
* protracted second stage of labour (more than two hours from full dilatation to delivery)
* more than 30 minutes of active pushing
* BMI > 35 kg/m2
* distance from skin to uterus > 8 cm
* age > 35 years old
* instrumental deliveries
* bleeding disorders
* polyhydramnios
* diabetes
* pre-eclampsia
* high blood pressure
* use of anticoagulant medications
* clinical chorioamnionitis
* placental abnormality (low-lying or abruption)
* fetal macrosomia
* uterine fibroids
* uterine anomalies
* previous uterine scar
* multiple pregnancy
* placental retention
* inability to follow procedures or insufficient knowledge of project language
* inability to give consent
* refusal to participate

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Women above 37 weeks of gestation without known risk factors for postpartum hemorrhage who have vaginal births in our centre will be eligible for this study
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Stiffness of the myometrium | Third labor stage to 30 minutes post placenta delivery
  Difference in median myometrial shear wave velocity between each time point: after fetal delivery, after placental delivery and 30 minutes after placental delivery.

SECONDARY OUTCOMES:
Blood loss | Two hours following the childbirth
  Measurement of total blood loss

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Lausanne, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided